CLINICAL TRIAL: NCT01124916
Title: Abdominal Colpopexy: Comparison of Endoscopic Surgical Strategies
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201805; RC1EB010649-01 (NIH)
Record Dates: First submitted 2010-05-06; First posted 2010-05-17 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Pelvic Organ Prolapse
Keywords: incontinence; prolapse; Abdominal sacrocolpopexy
MeSH Terms: conditions — Pelvic Organ Prolapse; Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic Abdominal Sacrocolpopexy (LASC) (Active Comparator): Women assigned to this cohort will receive standard laparoscopic abdominal sacrocolpopexy (LASC)
  Interventions: Procedure: Standard laparoscopic abdominal sacrocolpopexy
- Robotic Assisted Laparoscopic (RASC) (Experimental): Women assigned to this cohort will receive robotic assisted laparoscopic abdominal sacrocolpopexy (RASC)
  Interventions: Procedure: Robotic assisted laparoscopic abdominal sacrocolpopexy

INTERVENTIONS:
Procedure: Robotic assisted laparoscopic abdominal sacrocolpopexy — Robotic assisted laparoscopic abdominal sacrocolpopexy for surgical repair of pelvic organ prolapse.
  Other Names: RASC
  Arms: Robotic Assisted Laparoscopic (RASC)
Procedure: Standard laparoscopic abdominal sacrocolpopexy — Standard laparoscopic abdominal sacrocolpopexy for surgical repair of pelvic organ prolapse.
  Other Names: LASC
  Arms: Laparoscopic Abdominal Sacrocolpopexy (LASC)

SUMMARY:
The purpose of this research is to determine if there is a difference in total costs of care and return to health in women who undergo a laparoscopic abdominal sacrocolpopexy (ASC) compared to those undergoing the same procedure with the assistance of a robot.

Both traditional laparoscopic and robotic assisted laparoscopic approaches have been found to result in shorter hospital stays, decreased blood loss and similar surgical outcomes as compared to open abdominal surgery. The decision to use robotic assistance is typically based on surgeon preference and robot availability. The study will compare the outcomes of cost, quality of life, and return to work among women who undergo a laparoscopic sacrocolpopexy utilizing the robot to those using traditional laparoscopic techniques.

This research study is designed to compare the total costs and treatment success of these two surgical techniques. In addition, the study will compare outcomes of post-operative pain, quality of life, sexual function, return to normal activities and satisfaction with treatment outcome.

DETAILED DESCRIPTION:
Approximately one in ten women undergoes surgery for prolapse or incontinence in her lifetime. Of these, up to thirty percent require a re-operation for recurrence of their prolapse or incontinence symptoms. It has been estimated one in nine women will undergo a hysterectomy in her lifetime, and up to 10% of these women will require surgery for symptomatic vaginal vault prolapse. The search for the ideal repair for pelvic organ prolapse has led to the invention of several approaches to this problem.

Abdominal sacrocolpopexy (ASC) with synthetic mesh is considered the gold standard in the surgical management of pelvic organ prolapse with anatomic success rates ranging from 90 to 100%. Randomized comparative effectiveness trials and systematic literature reviews demonstrated the anatomic superiority of open ASC compared to vaginal sacrospinous ligament suspension.

Although ASC has the highest anatomic success rates for correcting apical prolapse, it is traditionally done via a laparotomy requiring an abdominal incision. Open technique is associated with more frequent short-term complications, including gastrointestinal.

Minimally invasive approaches to ASC using laparoscopy or robotic assisted laparoscopy demonstrate shorter hospital stays, decreased blood loss, and similar short-term anatomic outcomes when compared to open ASC. Increasing numbers of surgeons and patients choose minimally invasive ASC to maximize the benefits of abdominal placed mesh and the shorter-recovery associated with minimally invasive surgery. Few studies have compared laparoscopy to robotic assisted-laparoscopy in pelvic reconstructive surgery.

Like many techniques in pelvic surgery, trends in the management of pelvic organ prolapse continue to evolve. Unfortunately, such trends are not supported by robust data, specifically that provided by randomized clinical trials. Although robotic technology is new and rapidly spreading throughout the urologic and gynecologic communities, there are no randomized trials comparing outcomes of robotic to more traditional laparoscopic techniques for reconstructive pelvic surgery. Retrospective series indicate comparable efficacy with respect to cure of prolapse. However, to date is it unknown how robotic surgery compares to laparoscopic techniques with respect to cost, patient safety, pain, and ability to return to normal activities.

The use of the robot in laparoscopic surgery is costly. The costs of purchasing a robot has been estimated at $1.5 million dollars with annual maintenance costs of $112,0007. In addition, additional costs exist for the robotic equipment utilized with each case. It is arguable that the maintenance and operative equipment costs may overshadow any potential savings in length of hospital stay and patient convalescence. However, if robotic sacrocolpopexy can provide better immediate quality of life, less pain, and faster recovery compared to laparoscopic techniques, the investment in robotic techniques may very well be cost effective when a societal perspective is taken.

ELIGIBILITY:
Inclusion Criteria:

1. Stage II to IV pelvic organ prolapse
2. Prolapse of the vaginal apex or cervix to at least half way into the vaginal canal
3. Vaginal bulge symptoms
4. Minimally invasive surgery is planned
5. Available for 12 months of follow-up
6. Able to complete study assessments
7. Able and willing to provide written informed consent

Exclusion Criteria:

1. Contraindication to laparoscopic or robotically assisted laparoscopic abdominal sacrocolpopexy
2. Subject wishes to retain her uterus (i.e., surgical assignment may involve removal of uterus, if not previously removed)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kenton, M.D., Principal Investigator — Loyola University
Locations (2):
- United States (2):
  - UCLA, Los Angeles, California
  - Loyola University Medical Center, Maywood, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams P, Andersson KE, Birder L, Brubaker L, Cardozo L, Chapple C, Cottenden A, Davila W, de Ridder D, Dmochowski R, Drake M, Dubeau C, Fry C, Hanno P, Smith JH, Herschorn S, Hosker G, Kelleher C, Koelbl H, Khoury S, Madoff R, Milsom I, Moore K, Newman D, Nitti V, Norton C, Nygaard I, Payne C, Smith A, Staskin D, Tekgul S, Thuroff J, Tubaro A, Vodusek D, Wein A, Wyndaele JJ; Members of Committees; Fourth International Consultation on Incontinence. Fourth International Consultation on Incontinence Recommendations of the International Scientific Committee: Evaluation and treatment of urinary incontinence, pelvic organ prolapse, and fecal incontinence. Neurourol Urodyn. 2010;29(1):213-40. doi: 10.1002/nau.20870. No abstract available. PMID 20025020
- [Background] Nygaard IE, McCreery R, Brubaker L, Connolly A, Cundiff G, Weber AM, Zyczynski H; Pelvic Floor Disorders Network. Abdominal sacrocolpopexy: a comprehensive review. Obstet Gynecol. 2004 Oct;104(4):805-23. doi: 10.1097/01.AOG.0000139514.90897.07. PMID 15458906
- [Background] Benson JT, Lucente V, McClellan E. Vaginal versus abdominal reconstructive surgery for the treatment of pelvic support defects: a prospective randomized study with long-term outcome evaluation. Am J Obstet Gynecol. 1996 Dec;175(6):1418-21; discussion 1421-2. doi: 10.1016/s0002-9378(96)70084-4. PMID 8987919
- [Background] Maher CF, Qatawneh AM, Dwyer PL, Carey MP, Cornish A, Schluter PJ. Abdominal sacral colpopexy or vaginal sacrospinous colpopexy for vaginal vault prolapse: a prospective randomized study. Am J Obstet Gynecol. 2004 Jan;190(1):20-6. doi: 10.1016/j.ajog.2003.08.031. PMID 14749629
- [Background] McDermott CD, Hale DS. Abdominal, laparoscopic, and robotic surgery for pelvic organ prolapse. Obstet Gynecol Clin North Am. 2009 Sep;36(3):585-614. doi: 10.1016/j.ogc.2009.09.004. PMID 19932417
- [Background] Barbash GI, Glied SA. New technology and health care costs--the case of robot-assisted surgery. N Engl J Med. 2010 Aug 19;363(8):701-4. doi: 10.1056/NEJMp1006602. No abstract available. PMID 20818872
- [Background] Holtz DO, Miroshnichenko G, Finnegan MO, Chernick M, Dunton CJ. Endometrial cancer surgery costs: robot vs laparoscopy. J Minim Invasive Gynecol. 2010 Jul-Aug;17(4):500-3. doi: 10.1016/j.jmig.2010.03.012. Epub 2010 May 23. PMID 20547112
- [Background] Sarlos D, Kots L, Stevanovic N, Schaer G. Robotic hysterectomy versus conventional laparoscopic hysterectomy: outcome and cost analyses of a matched case-control study. Eur J Obstet Gynecol Reprod Biol. 2010 May;150(1):92-6. doi: 10.1016/j.ejogrb.2010.02.012. Epub 2010 Mar 5. PMID 20207063
- [Background] Paraiso MFR, Jelovsek JE, Frick A, Chen CCG, Barber MD. Laparoscopic compared with robotic sacrocolpopexy for vaginal prolapse: a randomized controlled trial. Obstet Gynecol. 2011 Nov;118(5):1005-1013. doi: 10.1097/AOG.0b013e318231537c. PMID 21979458
- [Background] Patel M, O'Sullivan D, Tulikangas PK. A comparison of costs for abdominal, laparoscopic, and robot-assisted sacral colpopexy. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Feb;20(2):223-8. doi: 10.1007/s00192-008-0744-2. Epub 2008 Oct 16. PMID 18923803
- [Background] Brink CA, Wells TJ, Sampselle CM, Taillie ER, Mayer R. A digital test for pelvic muscle strength in women with urinary incontinence. Nurs Res. 1994 Nov-Dec;43(6):352-6. PMID 7971299
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Shaw JW, Johnson JA, Coons SJ. US valuation of the EQ-5D health states: development and testing of the D1 valuation model. Med Care. 2005 Mar;43(3):203-20. doi: 10.1097/00005650-200503000-00003. PMID 15725977
- [Background] Barber MD, Walters MD, Cundiff GW; PESSRI Trial Group. Responsiveness of the Pelvic Floor Distress Inventory (PFDI) and Pelvic Floor Impact Questionnaire (PFIQ) in women undergoing vaginal surgery and pessary treatment for pelvic organ prolapse. Am J Obstet Gynecol. 2006 May;194(5):1492-8. doi: 10.1016/j.ajog.2006.01.076. PMID 16647933
- [Background] Rogers RG, Kammerer-Doak D, Villarreal A, Coates K, Qualls C. A new instrument to measure sexual function in women with urinary incontinence or pelvic organ prolapse. Am J Obstet Gynecol. 2001 Mar;184(4):552-8. doi: 10.1067/mob.2001.111100. PMID 11262452
- [Background] Hollenbeck BK, Dunn RL, Wolf JS Jr, Sanda MG, Wood DP, Gilbert SM, Weizer AZ, Montie JE, Wei JT. Development and validation of the convalescence and recovery evaluation (CARE) for measuring quality of life after surgery. Qual Life Res. 2008 Aug;17(6):915-26. doi: 10.1007/s11136-008-9366-x. Epub 2008 Jun 24. PMID 18574712
- [Background] Hedgepeth RC, Wolf JS Jr, Dunn RL, Wei JT, Hollenbeck BK. Patient-reported recovery after abdominal and pelvic surgery using the Convalescence and Recovery Evaluation (CARE): implications for measuring the impact of surgical processes of care and innovation. Surg Innov. 2009 Sep;16(3):243-8. doi: 10.1177/1553350609342075. Epub 2009 Aug 5. PMID 19661099
- [Background] Singer AJ, Arora B, Dagum A, Valentine S, Hollander JE. Development and validation of a novel scar evaluation scale. Plast Reconstr Surg. 2007 Dec;120(7):1892-1897. doi: 10.1097/01.prs.0000287275.15511.10. PMID 18090752
- [Background] Jelovsek JE, Barber MD. Women seeking treatment for advanced pelvic organ prolapse have decreased body image and quality of life. Am J Obstet Gynecol. 2006 May;194(5):1455-61. doi: 10.1016/j.ajog.2006.01.060. PMID 16647928
- [Background] Brubaker L, Cundiff GW, Fine P, Nygaard I, Richter HE, Visco AG, Zyczynski H, Brown MB, Weber AM; Pelvic Floor Disorders Network. Abdominal sacrocolpopexy with Burch colposuspension to reduce urinary stress incontinence. N Engl J Med. 2006 Apr 13;354(15):1557-66. doi: 10.1056/NEJMoa054208. PMID 16611949
- [Background] Richter HE, Albo ME, Zyczynski HM, Kenton K, Norton PA, Sirls LT, Kraus SR, Chai TC, Lemack GE, Dandreo KJ, Varner RE, Menefee S, Ghetti C, Brubaker L, Nygaard I, Khandwala S, Rozanski TA, Johnson H, Schaffer J, Stoddard AM, Holley RL, Nager CW, Moalli P, Mueller E, Arisco AM, Corton M, Tennstedt S, Chang TD, Gormley EA, Litman HJ; Urinary Incontinence Treatment Network. Retropubic versus transobturator midurethral slings for stress incontinence. N Engl J Med. 2010 Jun 3;362(22):2066-76. doi: 10.1056/NEJMoa0912658. Epub 2010 May 17. PMID 20479459
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Manca A, Hawkins N, Sculpher MJ. Estimating mean QALYs in trial-based cost-effectiveness analysis: the importance of controlling for baseline utility. Health Econ. 2005 May;14(5):487-96. doi: 10.1002/hec.944. PMID 15497198
- [Derived] Kenton K, Mueller ER, Tarney C, Bresee C, Anger JT. One-Year Outcomes After Minimally Invasive Sacrocolpopexy. Female Pelvic Med Reconstr Surg. 2016 Sep-Oct;22(5):382-4. doi: 10.1097/SPV.0000000000000300. PMID 27403758
- [Derived] Mueller ER, Kenton K, Anger JT, Bresee C, Tarnay C. Cosmetic Appearance of Port-site Scars 1 Year After Laparoscopic Versus Robotic Sacrocolpopexy: A Supplementary Study of the ACCESS Clinical Trial. J Minim Invasive Gynecol. 2016 Sep-Oct;23(6):917-21. doi: 10.1016/j.jmig.2016.05.001. Epub 2016 May 12. PMID 27180224
- [Derived] Anger JT, Mueller ER, Tarnay C, Smith B, Stroupe K, Rosenman A, Brubaker L, Bresee C, Kenton K. Robotic compared with laparoscopic sacrocolpopexy: a randomized controlled trial. Obstet Gynecol. 2014 Jan;123(1):5-12. doi: 10.1097/AOG.0000000000000006. PMID 24463657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from November 2009 to August 2011 (21 months)
Pre-assignment Details: Following enrollment, six women withdrew prior to randomization and two women were lost to follow-up prior to randomization
Period: Overall Study
Arm/Group | Laparoscopic Abdominal Sacrocolpopexy (LASC) | Robotic Assisted Laparoscopic (RASC)
Started | 38 | 40
Completed | 35 | 38
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprises all randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Laparoscopic Abdominal Sacrocolpopexy (LASC) | Robotic Assisted Laparoscopic (RASC) | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (9.2) | 58.5 (10.5) | 59.5 (9.9)
Gender [Count of Participants; unit: Participants]
  Female | 38 | 40 | 78
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 36 | 38 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 37 | 36 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
City and state where the study activities took place [Count of Participants; unit: Participants]
  Maywood, Illinois | 28 | 28 | 56
  Los Angeles, California | 10 | 12 | 22
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27 (4.7) | 28.2 (6.6) | 27.7 (5.7)
Parity [Mean (Standard Deviation); unit: Count of pregnancies] | 2.7 (1.3) | 2.6 (1.1) | 2.7 (1.2)
Years of Education [Count of Participants; unit: Participants]
  12 or fewer years | 14 | 14 | 28
  More than 12 years | 24 | 26 | 50
Net household income [Count of Participants; unit: Participants]
  Less than $50,000 | 18 | 11 | 29
  $50,000 to $75,000 | 11 | 11 | 22
  More than $75,000 | 8 | 15 | 23
  Unknown | 1 | 3 | 4
Comorbid Diabetes [Count of Participants; unit: Participants]
  No | 35 | 34 | 69
  Yes | 3 | 6 | 9
History of Heart Attack [Count of Participants; unit: Participants]
  No | 37 | 35 | 72
  Yes | 1 | 5 | 6
History of Stroke [Count of Participants; unit: Participants]
  No | 36 | 40 | 76
  Yes | 2 | 0 | 2
History of Cancer [Count of Participants; unit: Participants]
  No | 32 | 32 | 64
  Yes | 6 | 8 | 14
History of Stomach Ulcer [Count of Participants; unit: Participants]
  No | 31 | 30 | 61
  Yes | 7 | 10 | 17
Postmenopausal [Count of Participants; unit: Participants]
  No | 9 | 11 | 20
  Yes | 29 | 29 | 58
Concomitant estrogen therapy [Count of Participants; unit: Participants]
  No | 27 | 34 | 61
  Yes | 11 | 6 | 17
Previous surgery for urinary incontinence [Count of Participants; unit: Participants]
  No | 31 | 35 | 66
  Yes | 7 | 5 | 12
Previous surgery for pelvic organ prolapse [Count of Participants; unit: Participants]
  No | 30 | 32 | 62
  Yes | 8 | 8 | 16
Prior Hysterectomy [Count of Participants; unit: Participants]
  No | 19 | 26 | 45
  Yes | 19 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Total Cost of Care Between Standard and Robotic-assisted Laparoscopic Abdominal Sacrocolpopexy
Description: At 6-weeks following surgery, the study will measure the total cost of care in dollars and compare this estimate between women assigned to standard vs robotic-assisted laparoscopic abdominal sacrocolpopexy.
Time Frame: 6 Weeks
Population: The analysis for the primary outcome includes all randomized subjects.
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Laparoscopic Abdominal Sacrocolpopexy (LASC) | Robotic Assisted Laparoscopic (RASC)
Number analyzed (Participants) | 38 | 40
Dollars | 11573 (3191) | 19616 (3135)
Statistical Analysis 1: Comparison: Laparoscopic Abdominal Sacrocolpopexy (LASC) vs Robotic Assisted Laparoscopic (RASC); The null hypothesis is that there is no difference in the total cost of care between standard and robotic-assisted laparoscopic abdominal sacrocolpopexy six weeks after surgery; Test type: Superiority or Other; p < .001, t-test, 2 sided; Mean Difference (Net) = 8728, 95% CI 2-sided [7028.846 to 10427.154], Standard Error of Mean 853.129

2. Secondary Outcome: Urinary Distress Between Standard and Robotic-assisted Laparoscopic Abdominal Sacrocolpopexy
Description: At 6-months following surgery, the study will measure urinary distress using the Urinary Distress Inventory (UDI) and compare this estimate between women assigned to standard vs robotic-assisted laparoscopic abdominal sacrocolpopexy. The UDI measures urinary incontinence and distress and their effect on daily life. The score range is 0 to 300, with higher scores indicating worsening symptoms.
Time Frame: 6 Months
Population: The analysis excludes three individuals assigned to the LASC cohort and two individuals assigned to the RASC cohort because they were lost to follow-up six months after intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Laparoscopic Abdominal Sacrocolpopexy (LASC) | Robotic Assisted Laparoscopic (RASC)
Number analyzed (Participants) | 35 | 38
units on a scale | 25.1 (31.4) | 31.3 (35.3)
Statistical Analysis 1: Comparison: Laparoscopic Abdominal Sacrocolpopexy (LASC) vs Robotic Assisted Laparoscopic (RASC); The null hypothesis is that there is no difference in urinary distress between women assigned to LASC and those assigned to RASC six months after intervention as measured by the UDI; Test type: Superiority or Other; p = .43, t-test, 2 sided; Mean Difference (Net) = 6.20, 95% CI 2-sided [-21.769 to 9.369], Standard Error of Mean 7.846

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 1 year, 9 months
Arm/Group | Laparoscopic Abdominal Sacrocolpopexy (LASC) | Robotic Assisted Laparoscopic (RASC)
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 8/38 | 7/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laparoscopic Abdominal Sacrocolpopexy (LASC) (N=38) | Robotic Assisted Laparoscopic (RASC) (N=40)
Mesh Exposure (Surgical and medical procedures) | 0 (0) | 3 (3) — Suburethral Sling Mesh Exposure
Illiac Vein Injury (Surgical and medical procedures) | 1 (1) | 1 (1) — Left Iliac Vein Injury occurred at the time of the presacral dissection
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated Hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tissue granulation (Reproductive system and breast disorders) | 3 (4) | 0 (0) — Granulation of tissue was noted in the posterior midline of the vagina
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Mallory-Weiss tear (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (General disorders) | 0 (0) | 1 (1)
Intraoperative cystotomy (Surgical and medical procedures) | 1 (1) | 1 (1) — While passing the trocar, an Intraoperative Cystotomy was encountered. This was immediately identified by Cystoscopy and removed
Bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to specify.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No